CLINICAL TRIAL: NCT03347019
Title: Accelerated Rehabilitation After Arthroscopic Bankart Repair Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Irem Duzgun, associate professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 16/471-14
Record Dates: First submitted 2017-11-06; First posted 2017-11-20 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Bankart Lesion
Keywords: bankart repair; accelerated rehabilitation; shoulder
MeSH Terms: conditions — Bankart Lesions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- accelerated rehabilitation after surgery (Experimental): patients were included progressive rehabilitation programme first week after arthroscopic bankart repair consisting of passive shoulder range of motion exercises, scapular retraction exercises. The exercise programme progressed from active range of motion exercises to resistive and plyometric shoulder exercises. Patients were followed for six months.
  Interventions: Other: Accelerated rehabilitation
- delayed rehabilitation after surgery (Experimental): Patients were not allowed to start passive shoulder exercises first three weeks after surgery. Patients were included progressive rehabilitation programme third week after arthroscopic bankart repair consisting of passive shoulder range of motion exercises, scapular retraction exercises. The exercise programme progressed from active range of motion exercises to resistive and plyometric shoulder exercises. Patients were followed for six months.
  Interventions: Other: Delayed rehabilitation

INTERVENTIONS:
Other: Accelerated rehabilitation — advances in arthroscopic surgery have resulted in biomechanically stronger repairs that might allow for accelerated rehabilitation protocols and hence faster return to daily living activities and scapular control
  Arms: accelerated rehabilitation after surgery
Other: Delayed rehabilitation — Patients were not allowed to start rehabilitation programme first three weeks after surgery.
  Arms: delayed rehabilitation after surgery

SUMMARY:
The aim of this study was to prospectively evaluate the efficacy of an accelerated rehabilitation regime for patients undergoing early arthroscopic stabilization for first-time anterior dislocation in terms of clinical outcome, return to play data and recurrence rates.

DETAILED DESCRIPTION:
Traditional rehabilitation regimes post arthroscopic stabilization commonly stipulate a period of immobilization of between 2 weeks and 6 weeks.This is apparently embedded in practice and is reportedly based on tissue healing times. However early mobilisation would allow good clinical results in terms of clinical outcome, return to play data and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Patient were included based on their history of a clear mechanism of injury resulting in traumatic anterior dislocation, with clear evidence of labral injury confirmed on magnetic resonance imaging.

Exclusion Criteria:

* patients with inflammatory, autoimmune, endocrine or kidney diseases
* Recurrence
* Bony Bankart Lesion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
3 Dimensional Kinematic Analysis | at sixth months after surgery
  Scapular kinematic measurements were conducted by using three-dimensional electromagnetic system (Motion Monitor® Skeleton Analysis System, Innovative Sports Training Inc, Chicago, USA). The three-dimensional electromagnetic system consists of motion monitor software, transmitters and sensors integrated into this software (Flock of Birds System).

SECONDARY OUTCOMES:
Pain Assessment | at sixth months after surgery
  Pain was assessed by using numeric Visual Analogue Scale at rest, at night and during daily living activities. In numeric Visual Analogue Scale 0 represents "no pain", 10 represents "unbearable pain"
First Functional Assessment | at sixth months after surgery
  1. The Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities and that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms.This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.DASH Questionnaire will be calculated by using DASH Scoring Formula
Second Functional Assessment | at sixth months after surgery
  2. The American Shoulder and Elbow Surgeons Shoulder Score (ASES) is used to measure shoulder pain and functional limitations.The scores range from 0 to 100 and the highest score represents improvement in shoulder function after treatment interventions and to check the patient's ability to tolerate or perform the activities of daily living.
Third Functional Assessment | at sixth months after surgery
  3. Constant-Murley Shoulder Score (CONSTANT) is a 100-points scale composed of individual parameters.These parameters define the level of pain and the ability to carry out the normal daily activities of the patient.The Constant Score was introduced to determine the functionality after the treatment of a shoulder injury.The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion (40 points).The higher the score, the higher the quality of the function.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided